CLINICAL TRIAL: NCT05528302
Title: Technology Assisted and Remotely Delivered Cognitive Behavioural Therapy Intervention for Anxiety in People Living With Cognitive Impairment: Randomised Controlled Trial
Brief Title: Technology Assisted Cognitive Behavioural Therapy Intervention for Anxiety in People Living With Cognitive Impairment
Acronym: Tech-CBT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: Medical Research Future Fund (Other); Metro South Hospital and Health Services (Unknown); Metro North Hospital and Health Services (Unknown); Queensland University of Technology (Other); TalkVia (Unknown); Lions District 201Q3 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HREC/2022/QRBW/83925
Record Dates: First submitted 2022-07-19; First posted 2022-09-06 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Dementia; Cognitive Impairment; Anxiety
Keywords: Dementia; Cognitive Impairment; Anxiety; Cognitive Behavioural Therapy; Technology; Telehealth; Randomized Control Trial
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tech-CBT intervention (Experimental): Participants allocated to the Tech-CBT intervention group will attend six telehealth videoconferencing sessions - 1 session per week over 6 weeks. Each session will last between 60 to 90 minutes and will be facilitated by a trained therapist. During each session, the participant will learn and practice different psychotherapy techniques. The participant will be encouraged to practice these skills between sessions with the technology provided, either on their own or with the help of their support person.
  Interventions: Other: Tech-CBT intervention
- Control (No Intervention): Participants allocated to the Control group will receive usual care (i.e., no treatment for anxiety) and a mid-point check-in phone call/video call/email (depending on their preference) from the study team approximately 3 weeks after completing the initial questionnaires. This mid-point check-in is to identify whether there have been any changes to their usual care.

INTERVENTIONS:
Other: Tech-CBT intervention — The Tech-CBT intervention is a manualised package that incorporates Cognitive Behavioural Therapy methods.
  Arms: Tech-CBT intervention

SUMMARY:
This study is a randomized controlled trial (RCT) of a remotely-delivered, technology-assisted psychotherapy program, supported by an innovative software platform for people with cognitive impairment experiencing anxiety.

DETAILED DESCRIPTION:
Despite harmful health and economic consequences, anxiety is a vexing issue in persons with cognitive impairment with inadequate treatment options. What is needed currently is a digital technology option for treating anxiety in persons with cognitive impairment that can be rigorously evaluated and implemented. The objective of the study is to test the efficacy of a newly modified psychotherapy package (Tech-CBT), which incorporates Cognitive Behaviour Therapy (CBT) methods, assisted with technology and telehealth for persons with cognitive impairment experiencing anxiety. This project will also investigate the cost-effectiveness, usability and acceptability of Tech-CBT to enhance delivery of anxiety treatment for people with cognitive impairment. A process evaluation will inform its implementation in the community and memory clinics, and will recommend a strategic translational roadmap to enhance delivery of anxiety treatment in health services with a broad reach.

ELIGIBILITY:
Inclusion Criteria:

* Persons aged 18 years or over
* Persons with a diagnosis of mild cognitive impairment (MCI) or dementia of any aetiology based on a previous diagnosis by a clinician or scoring above threshold (≤32; MCI ≤32 and dementia ≤27) for cognitive impairment in the Modified Telephone Interview for Cognitive Impairment (TICS-M).
* Screening positive for anxiety (scoring ≥9 on Geriatric Anxiety Inventory, GAI), and/or subjective complaints of anxiety and/ or clinician diagnosis of a current anxiety disorder and screening positive for anxiety using the Rating Anxiety in Dementia scale (scoring ≥11 on RAID)

Exclusion Criteria:

* Persons with severe dementia
* Persons unable to communicate or complete questionnaires
* Persons who have a current risk of suicide within the last month as determined by the study clinical expert team.
* Persons with major depression as the primary complaint without reported symptoms of anxiety
* Persons with comorbid psychiatric conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-02-20 (Actual); Primary Completion 2025-10-22 (Actual); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Change in anxiety | Post-assessment (primary), 3 month follow-up and 6 month follow-up. Score ranging between 0 to 54 (lower score indicates better outcomes).
  Change from baseline in anxiety as measured by the Rating Anxiety in Dementia Scale (RAID).

SECONDARY OUTCOMES:
Change in quality of life | Post-assessment (~week 8), 3 month follow-up and 6 month follow-up. Score ranging between 0 to 52 (higher score indicates better outcomes).
  Change from baseline in quality of life as measured by the Quality of Life in Alzheimer's Disease (QoL-AD)
Change in anxiety | Post-assessment (~week 8), 3 month follow-up and 6 month follow-up. Score ranging between 0 to 20 (lower score indicates better outcomes).
  Change from baseline in anxiety as measured by the Geriatric Anxiety Inventory (GAI)
Change in worry | Post-assessment (~week 8), 3 month follow-up and 6 month follow-up. Score ranging between 8 to 40 (lower score indicates better outcomes).
  Change from baseline in worry as measured by the abbreviated version of the Penn State Worry Questionnaire (PSWQ-A).
Change in stress | Post-assessment (~week 8), 3 month follow-up and 6 month follow-up. Score ranging between 0 to 56 (lower score indicates better outcomes).
  Change from baseline in stress as measured by the Perceived Stress Scale (PSS-14).
Change in depressive symptoms | Post-assessment (~week 8), 3 month follow-up and 6 month follow-up. Score ranging between 0 to 15 (lower score indicates better outcomes).
  Change from baseline in depressive symptoms as measured by the Geriatric Depression Scale (GDS).
Change in carer burden | Post-assessment (~week 8), 3 month follow-up and 6 month follow-up. Score ranging between 0 to 88 (lower score indicates better outcomes).
  Change from baseline in carer burden as measured by the Zarit Burden Inventory (ZBI).
Change in carer quality of life | Post-assessment (~week 8), 3 month follow-up and 6 month follow-up. Score ranging between 20 to 99 (lower score indicates better outcomes).
  Change from baseline in carer quality of life as measured by the Assessment of Quality of Life (AQoL).
Change in carer depression and anxiety symptoms | Post-assessment (~week 8). Score ranging between 0 to 126 (lower score indicates better outcomes).
  Change from baseline in carer depression and anxiety symptoms as measured by the Depression Anxiety Stress Scales (DASS-21).
For people living with Parkinson's Disease, a change in Parkinsonism symptomology | Post-assessment (~week 8), 3 month follow-up and 6 month follow-up. Score ranging between 0 to 3500 (lower score indicates better outcomes).
  Change from baseline in Parkinsonism symptomology as measured by the Patient Reported Outcomes in Parkinson's Disease (PRO-PD).
For people living with Parkinson's Disease, a change in anxiety | Post-assessment (~week 8). Score ranging between 0 to 40 (lower score indicates better outcomes).
  Change from baseline in anxiety as measured by the Parkinson's disease Specific Anxiety Inventory (PDSAI).
For people living with Parkinson's Disease, a change in anxiety | Post-assessment (~week 8). Score ranging between 0 to 48 (lower score indicates better outcomes).
  Change from baseline in anxiety as measured by the Parkinson's Anxiety Scale (PAS).

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Queensland University of Technology, Brisbane, Queensland
  - Royal Brisbane and Women's Hospital (RBWH), Metro North Hospital and Health Services, Brisbane, Queensland
  - Surgical, Treatment and Rehabilitation Services (STARS), Metro North Hospital and Health Services, Brisbane, Queensland
  - The University of Queensland, Brisbane, Queensland
  - Princess Alexandra Hospital (PAH), Metro South Hospital and Health Services, Brisbane, Queensland

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) collected in this study will not be shared to other researchers.

REFERENCES:
- [Derived] Dissanayaka N, Brooks D, Worthy P, Mitchell L, Pachana NA, Byrne G, Keramat SA, Comans T, Bennett S, Liddle J, Chatfield MD, Broome A, Oram J, Appadurai K, Beattie E, Au T, King T, Welsh K, Pietsch A. A single-blind, parallel-group randomised trial of a Technology-assisted and remotely delivered Cognitive Behavioural Therapy intervention (Tech-CBT) versus usual care to reduce anxiety in people with mild cognitive impairment and dementia: study protocol for a randomised trial. Trials. 2023 Jun 20;24(1):420. doi: 10.1186/s13063-023-07381-2. PMID 37340492

DOCUMENTS (1):
  • Statistical Analysis Plan (2026-01-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT05528302/SAP_000.pdf